CLINICAL TRIAL: NCT05600075
Title: Microneedling With Topical Glycolic Acid 35% Versus Microneedling With Topical Insulin in the Treatment of Atrophic Post-acne Scars
Brief Title: Microneedling With Topical Preparations in the Treatment of Atrophic Post-acne Scars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Norhan Anees, Principal Investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: atrophic post-acne scars
Record Dates: First submitted 2022-10-21; First posted 2022-10-31 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Acne Scars - Mixed Atrophic and Hypertrophic
MeSH Terms: conditions — Hypertrophy | interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glycolic acid 35% group (Active Comparator): will be subjected to microneedling with topical glycolic acid 35%.
  Interventions: Drug: microneedling with topical glycolic acid 35%.
- topical insulin group (Active Comparator): will be subjected to microneedling with topical human insulin solution.
  Interventions: Drug: microneedling with topical human insulin solution.

INTERVENTIONS:
Drug: microneedling with topical glycolic acid 35%. — 15 patients will be subjected to microneedling with topical glycolic acid 35%. Selected patients will receive one session of microneedling combined with a topical agent, with two weeks interval till complete clearance or up to 6 sessions.
  Arms: Glycolic acid 35% group
Drug: microneedling with topical human insulin solution. — 15 patients will be subjected to microneedling with topical human insulin solution. Selected patients will receive one session of microneedling combined with a topical agent, with two weeks interval till complete clearance or up to 6 sessions.
  Arms: topical insulin group

SUMMARY:
To examine the anti-scarring effect of topical glycolic acid 35% combined with microneedling against that of topical insulin combined with microneedling for post acne scars

DETAILED DESCRIPTION:
Acne vulgaris (AV) is a common chronic inflammatory disease of skin that develops from sebaceous glands associated with hair follicles. Typically AV begins at puberty and may continue through adulthood affecting the comedogenic areas of face, back and chest .

One of the undesirable outcomes of acne is acne scars that are divided into two main types based on a loss (atrophic) or gain (hypertrophic) of collagen. Atrophic type is the most common type, further subdivided into three subtypes: icepick, boxcar and rolling scar .

Post acne scars occur in nearly 75% of patients with acne affecting both male and female equally . Acne scars impair quality of life and may be a risk factor for depression, suicide, low academic performance and unemployment .

There are different therapeutic modalities for atrophic acne scars including microneedling, chemical peeling, laser, filler, surgical procedures (punch excision, punch grafts) and fat transfer.

Microneedling is considered safe for all skin types. It is performed by dermapen or dermaroller to induce new collagen formation that remains for a few months after the procedure.

Microneedling enhances the effect of topical preparations when used combined with them due to increasing their absorption by creating small channels through the epidermis to the dermis .

It was reported that combination of glycolic acid (GA) with microneedling gave excellent results in treatment of post acne scars compared to microneedling alone.

Glycolic acid is an alpha hydroxy acid that decreases corneocytes cohesion leading to increasing keratinocytes turnover rate and faster desquamation .

It was found that glycolic acid increases dermal hyaluronic acid and collagen gene expression through increasing the secretion of IL6 .

the administration of topical human insulin was investigated for the treatment of atrophic post-acne scars and concluded that topical insulin following microneedling was associated with significant improvement.

Topical insulin induces collagen formation and neovascularization through synthesis of transforming growth factor (TGF b1) and vascular endothelial growth factor (VEGF).

ELIGIBILITY:
Inclusion Criteria:

* All types of facial atrophic acne scars
* Patients aged >18 years
* Both sexes

Exclusion Criteria:

* Pregnancy and lactation
* Active acne or any active facial lesion
* History of keloid scar
* History of systemic diseases as DM or hypotension
* Bleeding and coagulation disorders
* Infection and immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-22 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Goodman and Baron's acne scar grading system | through study completion, an average of 1 year
  Grade 1 Erythematous hypo or hyperpigmented flat marks Grade 2 Mild atrophy not obvious at social distance of >/=50 cm or easily covered by makeup or beard hair in male Grade 3 Moderate atrophy obvious at social distance of >/=50 cm, not easily covered by makeup or beard hair but able to be flattened by manual stretching of the skin Grade 4 Sever atrophy obvious at social distance >50 cm, not easily covered by makeup and not able to be flattened by manual stretching of skin
Quartile grading system | through study completion, an average of 1 year
  The improvement of patients is evaluated as follow:
  Poor (improvement < 25%) Mild (improvement 26%-50%) Good (improvement 51%-75%) Excellent (improvement >75%)
5 point scale for evaluating patient's satisfaction | through study completion, an average of 1 year
  None (no satisfaction) Mild (1%-25% satisfaction) Moderate (26%-50% satisfaction) Good (51%-75% satisfaction) Very good (76%-100% satisfaction)
Pain assessment | through study completion, an average of 1 year
  Pain during the session will be assessed and graded as mild, moderat and sever (Saadawi et al., 2018).

IPD SHARING:
Plan to Share IPD: Undecided